CLINICAL TRIAL: NCT05178251
Title: Impact of SARS-Cov2 Pandemic on Severity of Perioperative Complications in Patients Undergoing Appendectomy
Acronym: SAP-19
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Principal Investigator, Laurent BRUNAUD, Professor of Surgery, Central Hospital, Nancy, France
Other Study IDs: 2021PI185; 2021PI185 (Other: DRCI CHRU Nancy)
Record Dates: First submitted 2022-01-03; First posted 2022-01-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Complications; Appendicitis; COVID-19 Pandemic; Appendicitis With Peritonitis
Keywords: appendectomy; postoperative complications; covid 19
MeSH Terms: conditions — Postoperative Complications; Appendicitis; COVID-19 | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group without Covid 19 pandemic: - Patients who underwent an appendectomy from March 17, 2018 to December 14, 2018 and from March 17, 2019 to December 14, 2019
  Interventions: Procedure: appendectomy
- Test group with Covid 19 pandemic: - Patients who underwent an appendectomy from March 17, 2020 to December 14, 2020
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — appendectomy for acute appendicitis

SUMMARY:
There are 2 types of surgical procedures to remove the appendix : open appendectomy or laparoscopic appendectomy. About 60000 appendectomies are performed every year in France. Early diagnosis of acute appendicitis is essential to prevent the risk of disease progression, leading to complicated appendicitis and an increased risk for mortality. Data regarding appendicitis management in the literature are numerous. However, the impact of COVID-19 pandemic on the management of those patients has led to a decrease in the number of visits for acute appendicitis (ER), but a higher proportion of complicated appendicitis, probably due to the patient's delayed decision to go to emergency department at the onset of clinical symptoms. Complicated appendicitis may also lead to an overuse of antibiotics, a longer hospital stay, and a higher global cost for the health system. This aim of this study was to evaluate whether this hypothesis was valid for the regional NANCY-METZ area (CHR Metz and CHRU Nancy). The main research hypothesis was that the pandemic caused by SARS-COVID 19 was significantly linked to an increased incidence of perioperative complications in patients who underwent an appendectomy for acute appendicitis in this region (North-east part of France).

DETAILED DESCRIPTION:
Appendix is a finger-like, blind-ended tube connected to the cecum. The most frequent disease regarding the appendix is appendicitis. Appendicitis is an inflammation of the appendix caused by an obstruction of the lumen of the appendix. This obstruction is most commonly due to an appendicolith (calcified "stone" made of feces). Inflamed lymphoid tissue from a viral infection, parasites, gallstone, or tumors may also cause the blockage. This blockage leads to an increased pressure in the appendix, leading to a decreased blood flow to the tissues of the appendix, and bacterial growth inside the appendix causing inflammation. The combination of inflammation, reduced blood flow to the appendix and distention of the appendix causes tissue injury and lead to infection and potentially necrosis. If this process is left untreated, the appendix may burst, releasing bacteria into the abdominal cavity, leading to a peritonitis with a potential impact on mortality rate. Appendicitis symptoms include right lower abdominal pain, nausea, vomiting, and decreased appetite. Complicated appendicitis is defined as perforated appendicitis, peri-appendicular abscess or peritonitis. Consequently, acute appendicitis is considered to be a surgical emergency.

There are 2 types of surgical procedures to remove the appendix : open appendectomy or laparoscopic appendectomy. About 60000 appendectomies are performed every year in France. Early diagnosis of acute appendicitis is essential to prevent the risk of disease progression, leading to complicated appendicitis and an increased risk for mortality. Data regarding appendicitis management in the literature are numerous. However, the impact of COVID-19 pandemic on the management of those patients has led to a decrease in the number of visits for acute appendicitis (ER), but a higher proportion of complicated appendicitis, probably due to the patient's delayed decision to go to emergency department at the onset of clinical symptoms. Complicated appendicitis may also lead to an overuse of antibiotics, a longer hospital stay, and a higher global cost for the health system. This aim of this study was to evaluate whether this hypothesis was valid for the regional NANCY-METZ area (CHR Metz and CHRU Nancy). The main research hypothesis was that the pandemic caused by SARS-COVID 19 was significantly linked to an increased incidence of perioperative complications in patients who underwent an appendectomy for acute appendicitis in this region (North-east part of France).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent appendectomy

Exclusion Criteria:

* pregnancy
* protection of vulnerable adults
* disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed at :
  * CHR Mercy
  * CHRU nancy
  and who underwent appendectomy during the study period
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Perioperative complications after appendectomy | from March 17 to December 14 (2020-2021 versus 2019-2018)
  validated classification (Gomes classification)
Postoperative complications after appendectomy | from March 17 to December 14 (2020-2021 versus 2019-2018)
  validated classification (Clavien Dindo classification)

SECONDARY OUTCOMES:
Delay before surgery | from March 17 to December 14 (2020-2021 versus 2019-2018)
  Time duration from Symptoms onset and appendectomy
Hospitalization duration | from March 17 to December 14 (2020-2021 versus 2019-2018)
  Hospitalization duration
Antibiotherapy duration | from March 17 to December 14 (2020-2021 versus 2019-2018)
  Total antibiotherapy duration
Biological inflammatory syndrom | from March 17 to December 14 (2020-2021 versus 2019-2018)
  Hyperleucocytosis > 10000/mm3 and/or PCR > 100 mg/L
Type of hospitalisation | from March 17 to December 14 (2020-2021 versus 2019-2018)
  ward / ICU
Delay between appedectomy and postoperative complications | from March 17 to December 14 (2020-2021 versus 2019-2018)
  < 7 days; 7-30 days; > 30 days

CONTACTS AND LOCATIONS:
Overall Officials: laurent brunaud, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy - Département Chirurgie Viscérale, Métabolique et Cancérologique CVMC (7ème étage), Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhangu A; RIFT Study Group on behalf of the West Midlands Research Collaborative. Evaluation of appendicitis risk prediction models in adults with suspected appendicitis. Br J Surg. 2020 Jan;107(1):73-86. doi: 10.1002/bjs.11440. Epub 2019 Dec 3. PMID 31797357
- [Background] Gomes CA, Nunes TA, Fonseca Chebli JM, Junior CS, Gomes CC. Laparoscopy grading system of acute appendicitis: new insight for future trials. Surg Laparosc Endosc Percutan Tech. 2012 Oct;22(5):463-6. doi: 10.1097/SLE.0b013e318262edf1. PMID 23047394
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912